CLINICAL TRIAL: NCT04878783
Title: CT Scan-Based Radiomics and Molecular Expression Predictive Model to Assess Tumor Regression Grade Following Perioperative Chemotherapy in Esophago-Gastric Junction and Gastric Cancer
Brief Title: Radiomics and Molecular Expression Predictive Model for Esophago-Gastric Junction and Gastric Cancer TRG
Status: Active, not recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Andrea Laghi (Unknown)
Responsible Party: Principal Investigator, Giovanni Maria Garbarino, M.D., University of Roma La Sapienza
Other Study IDs: URomLS2022
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Adenocarcinoma of the Stomach
Keywords: radiomics; molecular expression; perioperative chemotherapy; FLOT; gastric cancer; esophago-gastric junction cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gastrectomy or esophagogastrectomy specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scan — Patients undergoing CT scan staging for gastric and EJ junction cancer + perioperative chemotherapy (FLOT regimen) , CT scan re-staging and radical gastrectomy or esophagogastrectomy will be enrolled in the study
  Other Names: FLOT chemotherapy; Radical Gastrectomy with D2 Lymphadenectomy; Radical Esophagogastrectomy with D2 Lymphadenectomy

SUMMARY:
The aim of this study is to develop a CT scan-based radiomics predictive model about tumor regression grade (TRG) in patients with esophago-gastric junction (EGJ) ang gastric cancer undergoing perioperative chemotherapy. The molecular expression of the neoplasms will be evaluated to assess its association with the TRG and the radiomic features.

DETAILED DESCRIPTION:
• To compare the radiomic features of the CT scans at the time of diagnosis (T0) and at the end of the preoperative chemotherapy (T1) in order to predict the TRG with the texture analysis on the first CT scan.

A non-good response (non-GR) has shown to be predictable with texture analysis on the pre-treatment CT scan.

Therefore, we hypothesize that texture analysis could let to identify the good response patients.

• To find correlation between the molecular expression of the tumor and the radiomics features.

Texture analysis on the pre-chemotherapy CT scan founded that entropy and compactness were higher and uniformity lower in responders. Nonetheless the association between radiomics features and molecular expression has not been investigated yet.

Therefore, we hypothesize to add some others radiomics signatures to the analysis and to find an association with the molecular expression.

• To find correlation between the molecular expression of the tumor and the TRG.

MSI gastric cancer has been shown to be less responsive to preoperative chemotherapy.

Therefore, we hypothesize to confirm this result.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven adenocarcinoma of the EGJ (Siewert II-III) or stomach.
* Preoperative staging: cT2-T4a, cN0-N3, M0.
* Patients >18 years old.
* Patients undergoing perioperative chemotherapy with Docetaxel, oxaliplatin, leucovorin, and 5-fluorouracil (FLOT).

Exclusion Criteria:

* Siewert I EGJ tumor
* Patients undergoing preoperative radiotherapy.
* Absence of both pre and post-chemotherapy CT-scan.
* Patients with tumor progression during preoperative chemotherapy.
* Patients undergoing other neoadjuvant chemotherapy regimen different from FLOT
* Exploratory laparoscopy with positive cytology on the peritoneal lavage or evidence of peritoneal carcinosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cT2-T4a, cN0-N3, M0 gastric or EGJ cancer who undergo FLOT perioperative chemotherapy followed by radical surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of radiomics analysis on the pre-treatment CT scan. | 2 months
  Comparing the radiomic features of the CT scans at the time of diagnosis (T0) and at the end of the preoperative chemotherapy (T1) in order to predict the TRG with the texture analysis on the first CT scan.

SECONDARY OUTCOMES:
Association of the radiomics features with the molecular expression of the tumor. | 2 months
  Texture analysis on the pre-chemotherapy CT scan founded that entropy and compactness were higher and uniformity lower in responders. Nonetheless the association between radiomics features and molecular expression has not been investigated yet.
  Therefore, we hypothesize to add some others radiomics signatures to the analysis and to find an association with the molecular expression.
Evaluation of the association between TRG and the molecular expression of the tumor. | 2 months
  Investigate if the molecular expression of the tumor can influence the TRG
Association between radiomics and molecular expression in regards to long-term outcomes | 5 years
  Analysis of the 3 and 5y DFS and OS of patients with the radiomics and molecular expression profile

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (4):
  - University of Padova, Padua
  - Link Campus University, Roma
  - Giovanni Maria Garbarino, Roma
  - University of Verona, Verona
- Amsterdam UMC location University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided